CLINICAL TRIAL: NCT00566033
Title: Multiple Intervention and AUdit in Renal Diseases to Optimize Care: the MAURO Study.
Brief Title: Multiple Intervention and AUdit in Renal Diseases to Optimize Care
Acronym: MAURO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy (Other Government)
Responsible Party: Principal Investigator, Carmine Zoccali, Prof., Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MAURO-001
Record Dates: First submitted 2007-11-29; First posted 2007-11-30 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Renal Insufficiency
Keywords: AUDIT; Chronic kidney disease; Clinical trial; Creatinine; Multiple intervents; Nephrology guidelines.
MeSH Terms: conditions — Renal Insufficiency; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: Audit-driven intervention
- 2 (No Intervention): Patients in this arm (arm 2) will undergo to standard care.

INTERVENTIONS:
Behavioral: Audit-driven intervention — Patients included in this arm will undergo to the multi-method quality improvement intervention (intensive intervention) that adds practice visits, telephone and e-mail contacts (for quality improvement facilitation) and audits to the approach of periodic guideline dissemination and feedback on demand used in the less intensive intervention.
  Arms: 1

SUMMARY:
Test whether the intensive intervention improves renal and cardiovascular outcomes in patients with chronic renal insufficiency.

Test whether a multi-method intensive intervention including clinical Audit improves adherence to a series of quality indicators relevant to hypertension control, proteinuria, treatment of dyslipidemia, anemia, calcium and phosphate alterations in patients with chronic renal insufficiency.

DETAILED DESCRIPTION:
Background:

Guidelines are currently promoted as a means for linking evidence based medicine to clinical practice and for reducing variation in clinical practice (1). However, there is ample evidence that implementation of evidence-based recommendations for prevention and management of renal disease progression and associated cardiovascular complications remain largely unsatisfactory (2). Deficiencies exist in the treatment of dyslipidemia and hypertension, inadequate use of angiotensin-converting enzyme inhibitors or angiotensin receptor blockers as well as in the treatment of anemia and of alterations in calcium and phosphate metabolism (2). Furthermore patients with diabetes mellitus infrequently receive recommended treatment for elevated glycosylated haemoglobin levels, hypertension, and dyslipidemia.

The importance of interventions to increase adherence to practice guidelines and to improve disease control is now widely perceived. However, little is known about the relative effectiveness of different implementation strategies. Fresh research is required to develop and validate practical strategies for improving the provision of evidence-based medicine in nephrology clinics. In particular, studies addressing multiple common, chronic conditions which simultaneously affect the population of patients with chronic renal insufficiency are now felt as of primary importance. The study was approved by Ethical Committees of all Nephrology Units participating into the MAURO study.

Specific hypotheses:

This study is designed as a clinical trial aimed at assessing whether a quality improvement intervention is more effective than standard care for improving adherence to a series of quality indicators relevant to the prevention of renal disease progression and associated cardiovascular complications. The multi-method quality improvement intervention (intensive intervention) adds telephone and e-mail contacts (for quality improvement facilitation) and audits to the approach of periodic guideline dissemination used in standard care.

Objective(s):

Test whether the intensive intervention improves renal and cardiovascular outcomes in patients with chronic renal insufficiency.

Test whether the intensive intervention improves adherence to a series of quality indicators relevant to hypertension control, proteinuria, treatment of dyslipidemia, anemia and calcium and phosphate alterations.

Endpoints:

The primary end point is a composite renal and cardiovascular end point, i.e. >30% decrease in the GFR, dialysis, transplantation, death or cardiovascular event [ECG documented angina or myocardial infarction, heart failure, arrhythmia (atrial fibrillation), cerebro-vascular event (stroke or transient ischemic attacks) or peripheral vascular diseases].

The renal unit-level outcome is the percentage of performance targets achieved. The patient level outcome is the percentage of patients for whom the recommended process measures occurs.

Key Inclusion Criteria:

* Average of at least 2 measurements of creatinine >1.5-4.0 mg/dL (males) and >1.3-3.5 mg/dL (females) during the six months run-in period or albuminuria> 30 mg/24h in at least two consecutive visits
* Previous diagnosis of specific nephropathy
* Non acute or rapidly evolving renal diseases
* Age range :18 - 75 years.
* Non-transplanted.
* Non-pregnant.
* Not affected by cancer or diseases in the terminal phase.

Study Design and procedures:

Randomized, controlled clinical trial, with the renal clinic as the unit of randomization.The two study arms (multi-intervention including AUDIT vs standard care) will be informed on the general aim of the study but will be kept blinded to the type of intervention made [(PRospective Blinded Intervention Design (PROBID)].

Drug Dosage, schedule and Route of Administration:

Drugs for the treatment of blood pressure, dyslipidemia, anemia and alterations in calcium phosphate metabolism will be administered according to doses recommended by the guidelines promoted by the Italian society of Nephrology and by the KDOQI guidelines.

Study duration:

Three years.

Sample Size for the primary end-point:

The sample size was calculated with the underlying assumption that the intracluster correlation coefficient (ICC)(estimated in a pilot study) be 0.016. The expected annual rate of the primary end point (at least 36% in 3 years) was derived from a previous study (3). With this background in mind, we found that allocating 330 patients in the active arm and 330 in the control arm, the study will have a 80% power for capturing as statistically significant (P <0.05, two tailed) a 1/3 risk reduction in three years (36% vs 24%) in the intensive intervention group.

Corollary information:

During the study a sera and DNA data-bank will be created to allow testing a series of open questions on renal disease progression and associated cardiovascular complications.

Ethical considerations:

The protocol is in conformity with the declaration of Helsinki and informed consent will be asked for to all participants.

Nephrology Units participating into the MAURO study:

Reggio Calabria, Melito(RC), Locri(RC), Palmi(RC), Taurianova(RC), Catanzaro(2 Units), Soverato(CZ), Lamezia(CZ), Cosenza, Lungro(CS), Rossano(CS), S.Giovanni in Fiore(CS), Paola(CS), Amantea-Praia a Mare(CS), Vibo Valentia-Tropea-Soriano(VV), Crotone, Messina, Catania, Acireale(CT), Sassari, Francavilla(TA).

References:

1. Hayward RS. Clinical practice guidelines on trial. CMAJ 1997; 156:1725-1727.
2. De Nicola L, Minutolo R, Chiodini P, Zoccali C, Castellino P, Donadio C, Strippoli M, Casino F, Giannattasio M, Petrarulo F, Virgilio M, Laraia E, Di Iorio BR, Savica V, Conte G; TArget Blood Pressure LEvels in Chronic Kidney Disease (TABLE in CKD) Study Group. Global approach to cardiovascular risk in chronic kidney disease: reality and opportunities for intervention. Kidney Int 2006;69:538-545.
3. Sarnak MJ, Greene T, Wang X, Beck G, Kusek JW, Collins AJ, Levey AS.The effect of a lower target blood pressure on the progression of kidney disease: long-term follow-up of the modification of diet in renal disease study.1: Ann Intern Med 2005; 142: 342-351.

ELIGIBILITY:
Inclusion Criteria:

* Creatinine >1.5 -4.0 mg/dL (males) and >1.3-3.5 mg/dL (females).
* Age range :18 - 75 years

Exclusion Criteria:

* Transplanted
* Pregnant
* Affected by cancer or diseases in the terminal phase
* Non acute or rapidly evolving renal diseases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 788 (Actual)
Dates: Start 2006-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
A composite renal and cardiovascular (CV) end point, i.e. >30% decrease in the GFR, dialysis, transplantation, death or CV event. | 3 years

SECONDARY OUTCOMES:
The primary renal unit-level outcome is the percentage of performance targets achieved. The primary patient-level outcome is the percentage of patients for whom the recommended process measures occurs. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Carmine Zoccali, Prof., Study Director — CNR-IBIM & Nephrology Unit of Reggio Calabria
Locations (1):
- Nephrology Units participating to the MAURO study in the, Calabrian, Sicily, Puglia and Sardenia Regions, Italy

REFERENCES:
- [Background] Hayward RS. Clinical practice guidelines on trial. CMAJ. 1997 Jun 15;156(12):1725-7. No abstract available. PMID 9220924
- [Background] De Nicola L, Minutolo R, Chiodini P, Zoccali C, Castellino P, Donadio C, Strippoli M, Casino F, Giannattasio M, Petrarulo F, Virgilio M, Laraia E, Di Iorio BR, Savica V, Conte G; TArget Blood Pressure LEvels in Chronic Kidney Disease (TABLE in CKD) Study Group. Global approach to cardiovascular risk in chronic kidney disease: reality and opportunities for intervention. Kidney Int. 2006 Feb;69(3):538-45. doi: 10.1038/sj.ki.5000085. PMID 16395261
- [Background] Kerry SM, Bland JM. The intracluster correlation coefficient in cluster randomisation. BMJ. 1998 May 9;316(7142):1455. doi: 10.1136/bmj.316.7142.1455. No abstract available. PMID 9572764
- [Derived] Leonardis D, Mallamaci F, Enia G, Postorino M, Tripepi G, Zoccali C; MAURO Study Investigators. The MAURO study: baseline characteristics and compliance with guidelines targets. J Nephrol. 2012 Nov-Dec;25(6):1081-90. doi: 10.5301/jn.5000239. PMID 23172127